CLINICAL TRIAL: NCT02130336
Title: The Effects of High-intensity Aerobic Training in Patients With Metabolic Syndrome and Its Dose Response Study
Brief Title: The Effects of High-intensity Aerobic Training in Patients With Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 201112105RIC
Record Dates: First submitted 2014-04-28; First posted 2014-05-05 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Metabolic Syndrome X; Exercise; Physical Activity
Keywords: Metabolic syndrome; Metabolic risk factors; High-intensity interval training; Moderate-intensity exercise
MeSH Terms: conditions — Metabolic Syndrome; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aerobic interval training (Experimental): Frequency: Exercise 3 times a week. Twice under supervision and home exercise once a week.
  Duration: Totally 40 minutes in one session. Intensity: 10-minute warm-up and 5-minute cool-down at 40% maximal heart rate (HRmax), participants and exercise 4-minute high-intensity training at 85-90% HRmax and 4 times separated by 3-minute active recovery at 70% HRmax.
  Type: Using treadmill while under supervision.
  Interventions: Behavioral: Aerobic interval training
- Continuous moderate-intensity exercise (Experimental): Frequency: 5 times a week. Twice under supervision and home exercise 3 times a week.
  Duration: Totally 45 minutes per session. Intensity: 10-minute warm-up at 40% maximal heart rate (HRmax), 30-minute moderate intensity exercise at 50-70% HRmax and 5-minute cool-down at 40% HRmax Type: Using treadmill under supervision.
  Interventions: Behavioral: Continuous moderate-intensity exercise
- Control group (No Intervention): Subjects in control group will receive general exercise knowledge and counseling.

INTERVENTIONS:
Behavioral: Aerobic interval training
  Other Names: AIT; High-intensity interval training
  Arms: Aerobic interval training
Behavioral: Continuous moderate-intensity exercise
  Other Names: CME; Continuous moderate-intensity training
  Arms: Continuous moderate-intensity exercise

SUMMARY:
Background. The prevalence of metabolic syndrome (MetS) has been increasing, and its risk is positively correlated with age. Due to ageing society in Taiwan, how to treat metabolic syndrome and decrease the complications is an important health issue. Relatively few studies have been focusing on the effects of exercise training in patients with MetS with long-term follow-up. Recently, high-intensity interval training or aerobic interval training (AIT) consisting of high intensity separated by active recovery has been proposed to be more effective than isocaloric continuous moderate-intensity exercise (CME) in raising exercise capacity (VO2max) in some specific patient population.

Purpose. The purposes are to (1) compare the effects of 16-week CME and AIT on reducing the numbers of metabolic risk factors in patients with MetS and the prevalence.

Hypothesis: 16-week AIT reduces more metabolic risk factors than CME in patients with MetS.

Methods. This study will be a multiple-center trial. One hundred and twenty patients, aged ≥45 years, with a diagnosis of MetS for each center will be recruited. Subjects will be randomly assigned to either control, CME, or AIT group after baseline assessments. Participants in control group will receive usual care and the others in two exercise groups will undergo 16-week exercise training. All subjects will receive 16-week, 6-month and 1-year follow-ups including blood test, body composition (body mass index, waist circumference), pulse wave velocity, and maximal exercise testing. Statistical analysis will be conducted using SPSS 11.5, p < 0.05 indicating statistical significance. Data will be presented in mean±standard deviation or number (percentile) with intention-to-treat analysis. Chi-square test or one-way Analysis of Variance (ANOVA) will be used to compare whether there are between-group differences at baseline. Two-way repeated measures ANOVA and post-hoc test will be performed to examine time and group effect if there is interaction effect, otherwise Bonferroni will be used. The subgroup analysis between MetS and n-MetS after training will be performed using the same statistical methods.

DETAILED DESCRIPTION:
Intervention (exercise) protocol:

1. CME group: exercise at least 30-minute moderate intensity 5 times a week, twice on treadmill under supervision and home exercise 3 times a week. CME protocol including 10-minute warm-up at 40% maximal heart rate (HRmax), 30-minute moderate intensity exercise at 50-70% HRmax and 5-minute cool-down at 40% HRmax
2. AIT group: exercise 3 times a week including twice on treadmill under supervision and home exercise once a week. AIT protocol including 10-minute warm-up and 5-minute cool-down at 40% HRmax, participants and exercise 4-minute high-intensity training at 85-90% HRmax and 4 times separated by 3-minute active recovery at 70% HRmax.

ELIGIBILITY:
Inclusion Criteria:

* 45-75 years old
* diagnosis of metabolic syndrome
* able to follow the instruction

Exclusion Criteria:

* unstable hypertension
* coronary artery disease or pulmonary diseases
* chronic kidney failure
* unable to perform exercise

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-05 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in metabolic risk factors at 16-week | baseline and 16-week
  Using blood test and anthropometric measurement to examine the differences between time points.
Change from baseline in metabolic risk factors at 6-month follow-up | baseline and 6-month after intervention completed
  Using blood test and anthropometric measurement to examine the differences between time points.
Change from baseline in metabolic risk factors at 1-year follow-up | baseline and 1-year after intervention completed
  Using blood test and anthropometric measurement to examine the differences between time points.

SECONDARY OUTCOMES:
Change from baseline in exercise capacity at 16-week | baseline and 16-week
  Using exercise testing to evaluate peak oxygen consumption at peak exercise to know the cardiopulmonary fitness in all subjects.
Change from baseline in heart rate variability at 16-week | baseline and 16-week
  Assessing continuous heart rate at resting (10-min), during exercise testing, and after exercise testing (10-min) and further analyzing heart rate variability in time and frequency domain.
Change from baseline in pulse wave velocity at 16-week | baseline and 16-week
  Assessing blood pressure in four limbs to analyze pulse wave velocity and evaluate the stiffness of peripheral arteries.
Change from baseline in level of physical activity at 16-week | baseline and 16-week
  Using 7-day recall physical activity questionnaire to examine the level of physical activity.
Change from baseline in dietary status at 16-week | baseline and 16-week
  Using dietary log to calculate caloric intake in recent one day.
Change from baseline in metabonomics at 16-week | baseline and 16-week
  Using blood test to analyze the differences in the activity of metabonomics.
Change from baseline in exercise capacity at 6-month follow-up | baseline and 6-month after intervention completed
  Using exercise testing to evaluate peak oxygen consumption at peak exercise to know the cardiopulmonary fitness in all subjects.
Change from baseline in exercise capacity at 1-year follow-up | baseline and 1-year after intervention completed
  Using exercise testing to evaluate peak oxygen consumption at peak exercise to know the cardiopulmonary fitness in all subjects.
Change from baseline in heart rate variability at 6-month follow-up | baseline and 6-month after intervention completed
  Assessing continuous heart rate at resting (10-min), during exercise testing, and after exercise testing (10-min) and further analyzing heart rate variability in time and frequency domain.
Change from baseline in heart rate variability at 1-year follow-up | baseline and 1-year after intervention completed
  Assessing continuous heart rate at resting (10-min), during exercise testing, and after exercise testing (10-min) and further analyzing heart rate variability in time and frequency domain.
Change from baseline in pulse wave velocity at 6-month follow-up | baseline and 6-month after intervention completed
  Assessing blood pressure in four limbs to analyze pulse wave velocity and evaluate the stiffness of peripheral arteries.
Change from baseline in pulse wave velocity at 1-year follow-up | baseline and 1-year after intervention completed
  Assessing blood pressure in four limbs to analyze pulse wave velocity and evaluate the stiffness of peripheral arteries.
Change from baseline in level of physical activity at 6-month follow-up | baseline and 6-month after intervention completed
  Using 7-day recall physical activity questionnaire to examine the level of physical activity.
Change from baseline in level of physical activity at 1-year follow-up | baseline and 1-year after intervention completed
  Using 7-day recall physical activity questionnaire to examine the level of physical activity.
Change from baseline in dietary status at 6-month follow-up | baseline and 6-month after intervention completed
  Using dietary log to calculate caloric intake in recent one day.
Change from baseline in dietary status at 1-year follow-up | baseline and 1-year after intervention completed
  Using dietary log to calculate caloric intake in recent one day.
Change from baseline in metabonomics at 6-month follow-up | baseline and 6-month after intervention completed
  Using blood test to analyze the differences in the activity of metabonomics.
Change from baseline in metabonomics at 1-year follow-up | baseline and 1-year after intervention completed
  Using blood test to analyze the differences in the activity of metabonomics.

CONTACTS AND LOCATIONS:
Overall Officials: Meng-Yueh Chien, Ph.D, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan